CLINICAL TRIAL: NCT02136017
Title: Phase 4 Study of Post-License Safety Evaluation of Influenza Split Vaccine
Brief Title: Post-License Safety Evaluation of Influenza Virus Vaccine
Status: Completed | Type: Observational
Sponsor: Sichuan Center for Disease Control and Prevention (Other Government)
Collaborators: China National Biotec Group Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: cnbg-002
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Influenza; Adverse Drug Event
Keywords: AEFI; influenza vaccine
MeSH Terms: conditions — Influenza, Human; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Changchun biologial's vaccine: Changchun Biological's vaccine group is the population injected with this vaccine.

SUMMARY:
To evaluate the safety of the post-licensed influenza virus vaccine made of Changchun Institute of Biological Products Co.,Ltd.

DETAILED DESCRIPTION:
In order to evaluate the safety of the post-licensed influenza vaccine (the vaccine is manufactured by Changchun Institute of Biological Products Co.,Ltd in China), retrospectively collect the AEFI cases reported from national AEFI surveillance system in Sichuan province of China in 2013, compare the incidence and proportion of local and general reactions, with other influenza vaccine.

Adverse events were collected through the National Immunization Information System's National Adverse Events Following Immunization (AEFI) Surveillance System, which was established in 2005 on the basis of World Health Organization (WHO) guidelines. According to the Guideline for the Identification of Adverse Reaction after Immunization issued by the Chinese Ministry of Health in 2008, Sichuan CDC and local prefectural CDC must organize an expert panel to investigate adverse events and assess causality, using criteria based on Chinese Standard Procedures for Vaccination.

At the time of vaccination, vaccinees were instructed to report any adverse event to physicians or vaccination providers. Adverse events that were fatal or that resulted in disability and clusters of events (i.e., notably high numbers of similar adverse events related to a certain vaccine) were required to be reported within 2 hours after their occurrence. The following adverse events were required to be reported within 2 days after their occurrence: anaphylaxis or other allergic reactions occurring within 24 hours after vaccination; fever (axillary temperature, >37.5°C), angioedema, or a local injection-site reaction (diameter, >2.5 cm) occurring within 5 days after vaccination; purpura, an Arthus reaction, febrile convulsion, seizure, or polyneuritis occurring within 15 days after vaccination; and the Guillain-Barré syndrome occurring within 3 months after vaccination. Other reactions that were common and minor (e.g., mild pain and fatigue) were not required to be reported.

ELIGIBILITY:
Inclusion Criteria:

* ever vaccinated one dose influenza vaccine(manufactured by Changchun institute of biological product) in 2013
* above 3 years old

Exclusion Criteria:

* Severe allergic reaction (e.g., anaphylaxis) after previous dose of any IIV or LAIV
* allergic to a vaccine component, including egg protein.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all the people immunized by influenza vaccine of Changchun Institute of Biological Product in Sichuan province in 2013.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
occurence rate of adverse reaction | 1 month after vaccination
  the general or local reactions are reported after vaccination .

CONTACTS AND LOCATIONS:
Overall Officials: rui ao, master, Principal Investigator — Sichuan CDC